CLINICAL TRIAL: NCT04653974
Title: Comparative Evaluation of Pain Perception With a New Needle-Free System and Dental Injection in Children: A Randomized Clinical Trial
Brief Title: Pain Perception of Needle-free System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halenur Altan, Associated Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1257-5993
Record Dates: First submitted 2020-11-28; First posted 2020-12-04 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Pain; Needle Phobia; Anxiety; Dental Fear; Local Anesthesia
Keywords: Children; Dental injection; Needle-free injection system; Pain; Pulpotomy
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Dental Health Services

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needle-free injection group (Active Comparator): In needle-free injection techniques, 2% lidocaine with 1/80.000 epinephrine (Lidocaine, Colombia) was injected using the Comfort-In system.
  Interventions: Behavioral: Needle-free injection
- Dental injection group (Active Comparator): In the conventional dental-injection method, 2% lidocaine with 1/80.000 epinephrine (Lidocaine, Colombia) was injected using a 27G, 40-mm, disposable syringe with a needle.
  Interventions: Behavioral: Needle-free injection

INTERVENTIONS:
Behavioral: Needle-free injection — This study was performed among children aged 4-11 years who required dental treatment and were treated at the Department of Pedodontics, Faculty of Dentistry, Gaziosmanpasa University. A total of 70 patients were evaluated in accordance with the exclusion criteria and 56 children (31 girls and 25 boys) were included in this study. Children who needed dental treatment were randomly divided into two groups. All dental injections were administered by the same operator (MB), a pediatric dentist with two years of experience in using the Comfort-In system.
  In both groups, the children were asked to rate their pain intensity by choosing the closest statement on the Wong-Baker Pain Scale at three time points: immediately after injection (Pain 1), during treatment (Pain 2), and at the end of the treatment (Pain 3).
  Other Names: Dental injection

SUMMARY:
The purpose of this study is to evaluate and compare the pain perception associated with a needle-free injection system( Comfort-In) and dental injection method in filling and pulpotomy treatments

DETAILED DESCRIPTION:
Needle-free injection system(Comfort-In) and dental injection method was applied on the teeth of children who need dental treatment.70 patients were included in the study. Patients were randomized into two grups according to the injection technique.

Group1: Needle-free injection system(Comofrt-In) 2:Dental injection method. The pain intensity was assessed during anesthesia, during treatment and at the end of thetreatment by the Wong Baker Faces Pain Scale.

The datas were analyzed with a three-way variance method in repeated.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 4-11 years
* Having no developmental or systemic disorder or no history of allergy
* Having "positive" or "definitely positive" cooperation level according to the Frankl Behavior Scale
* Having sufficient mouth opening
* Operation only on primary teeth
* Having decayed teeth that require anesthesia

Exclusion Criteria:

* Patients younger than five years, older than 11 years,
* Patients with systemic or developmental disorders
* Children with an allergy history
* 'Negative' or 'definitly negative' behavior rating according to the Frankl scale
* Patients whose mouth opening is not sufficient for dental treatment
* Operating only on permanent teeth
* Teeth that are beyond the treatment stage
* When pain occurred during treatment, supplemental anesthetics administrated, and these children were excluded.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Pain at different anesthesia methods | after dental treatments to 24 hour
  The pain perception scores in the two anesthesia methods were assessed with Wong-Baker Pain Scale (Wong-Baker Scale is pain assessment method.It consists of 6 facial expressions that are evaluated from 0 to 10 according to the severity of the pain.)

CONTACTS AND LOCATIONS:
Overall Officials: Halenur Altan, Assoc Prof., Principal Investigator — Tokat Gaziosmanpasa University, Faculty of Dentistry, Department of Pediatric Dentistry
Locations (1):
- Tokat Gaziosmanpasa University, Faculty of Dentistry, Tokat Province, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makade CS, Shenoi PR, Gunwal MK. Comparison of acceptance, preference and efficacy between pressure anesthesia and classical needle infiltration anesthesia for dental restorative procedures in adult patients. J Conserv Dent. 2014 Mar;17(2):169-74. doi: 10.4103/0972-0707.128063. PMID 24778516
- [Background] Arapostathis KN, Dabarakis NN, Coolidge T, Tsirlis A, Kotsanos N. Comparison of acceptance, preference, and efficacy between jet injection INJEX and local infiltration anesthesia in 6 to 11 year old dental patients. Anesth Prog. 2010 Spring;57(1):3-12. doi: 10.2344/0003-3006-57.1.3. PMID 20331333
- [Background] Oliveira ACA, Amorim KS, Nascimento Junior EMD, Duarte ACB, Groppo FC, Takeshita WM, Souza LMA. Assessment of anesthetic properties and pain during needleless jet injection anesthesia: a randomized clinical trial. J Appl Oral Sci. 2019 Jan 14;27:e20180195. doi: 10.1590/1678-7757-2018-0195. PMID 30673030
- [Background] Greenfield W, Karpinski JF. Clinical application of jet injection to comprehensive pain control. Anesth Prog. 1973 Jul-Aug;20(4):110-2. No abstract available. PMID 4516579
- [Background] Saravia ME, Bush JP. The needleless syringe: efficacy of anesthesia and patient preference in child dental patients. J Clin Pediatr Dent. 1991 Winter;15(2):109-12. PMID 1931745
- [Background] Baghlaf K, Alamoudi N, Elashiry E, Farsi N, El Derwi DA, Abdullah AM. The pain-related behavior and pain perception associated with computerized anesthesia in pulpotomies of mandibular primary molars: A randomized controlled trial. Quintessence Int. 2015 Oct;46(9):799-806. doi: 10.3290/j.qi.a34553. PMID 26287025
- [Background] Munshi AK, Hegde A, Bashir N. Clinical evaluation of the efficacy of anesthesia and patient preference using the needle-less jet syringe in pediatric dental practice. J Clin Pediatr Dent. 2001 Winter;25(2):131-6. doi: 10.17796/jcpd.25.2.q6426p853266q575. PMID 11314212
- [Background] Ogle OE, Mahjoubi G. Advances in local anesthesia in dentistry. Dent Clin North Am. 2011 Jul;55(3):481-99, viii. doi: 10.1016/j.cden.2011.02.007. PMID 21726685
- [Background] Sermet Elbay U, Elbay M, Yildirim S, Kaya E, Kaya C, Ugurluel C, BaydemIr C. Evaluation of the injection pain with the use of DentalVibe injection system during supraperiosteal anaesthesia in children: a randomised clinical trial. Int J Paediatr Dent. 2016 Sep;26(5):336-45. doi: 10.1111/ipd.12204. Epub 2015 Sep 15. PMID 26369274
- [Background] Oztas N, Olmez A, Yel B. Clinical evaluation of transcutaneous electronic nerve stimulation for pain control during tooth preparation. Quintessence Int. 1997 Sep;28(9):603-8. PMID 9477875
- [Background] Goodell GG, Gallagher FJ, Nicoll BK. Comparison of a controlled injection pressure system with a conventional technique. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2000 Jul;90(1):88-94. doi: 10.1067/moe.2000.107365. PMID 10884642
- [Background] Gibson RS, Allen K, Hutfless S, Beiraghi S. The Wand vs. traditional injection: a comparison of pain related behaviors. Pediatr Dent. 2000 Nov-Dec;22(6):458-62. PMID 11132503
- [Background] Asarch T, Allen K, Petersen B, Beiraghi S. Efficacy of a computerized local anesthesia device in pediatric dentistry. Pediatr Dent. 1999 Nov-Dec;21(7):421-4. PMID 10633514
- [Background] Ocak H, Akkoyun EF, Colpak HA, Demetoglu U, Yucesoy T, Kilic E, Alkan A. Is the jet injection effective for teeth extraction? J Stomatol Oral Maxillofac Surg. 2020 Feb;121(1):19-24. doi: 10.1016/j.jormas.2019.05.001. Epub 2019 May 8. PMID 31077857
- [Background] Kuensting LL, DeBoer S, Holleran R, Shultz BL, Steinmann RA, Venella J. Difficult venous access in children: taking control. J Emerg Nurs. 2009 Sep;35(5):419-24. doi: 10.1016/j.jen.2009.01.014. Epub 2009 Mar 21. No abstract available. PMID 19748021
- [Background] Milgrom P, Coldwell SE, Getz T, Weinstein P, Ramsay DS. Four dimensions of fear of dental injections. J Am Dent Assoc. 1997 Jun;128(6):756-66. doi: 10.14219/jada.archive.1997.0301. PMID 9188235
- [Background] Splieth CH, Bunger B, Pine C. Barriers for dental treatment of primary teeth in East and West Germany. Int J Paediatr Dent. 2009 Mar;19(2):84-90. doi: 10.1111/j.1365-263X.2008.00949.x. Epub 2008 Dec 19. PMID 19207736
- [Background] Oosterink FM, de Jongh A, Aartman IH. What are people afraid of during dental treatment? Anxiety-provoking capacity of 67 stimuli characteristic of the dental setting. Eur J Oral Sci. 2008 Feb;116(1):44-51. doi: 10.1111/j.1600-0722.2007.00500.x. PMID 18186731
- [Background] Deepak V, Challa RR, Kamatham R, Nuvvula S. Comparison of a New Auto-controlled Injection System with Traditional Syringe for Mandibular Infiltrations in Children: A Randomized Clinical Trial. Anesth Essays Res. 2017 Apr-Jun;11(2):431-438. doi: 10.4103/0259-1162.194535. PMID 28663636
- [Derived] Altan H, Belevcikli M, Cosgun A, Demir O. Comparative evaluation of pain perception with a new needle-free system and dental needle method in children: a randomized clinical trial. BMC Anesthesiol. 2021 Dec 1;21(1):301. doi: 10.1186/s12871-021-01524-1. PMID 34852779